CLINICAL TRIAL: NCT03478917
Title: Studies to Facilitate the Early Diagnosis of Sickle Acute Chest Syndrome Using a Combination of Plasma Biomarkers and Chest Imaging
Brief Title: Early Diagnosis of Sickle Acute Chest Syndrome Using a Combination of Plasma Bimarkers and Chest Imaging
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999918065; 18-H-N065
Record Dates: First submitted 2018-03-23; First posted 2018-03-27 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07-13

CONDITIONS: Sickle Cell Disease (SCD)
Keywords: Vasoocclusive Crisis (VOC); Sickle Cell Disease (SCD); Acute Chest Syndrome (ACS); Pulmonary Syndrome; Pneumonia; Natural History
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises; Acute Chest Syndrome; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arm 1: Subjects previously enrolled onto protocol 05-H-0019 who were hospitalized with vasoocclusivecrisis.

SUMMARY:
Background:

Painful vasoocclusive crisis (VOC) occurs in people with sickle cell disease (SCD). People with VOC have many visits to the hospital. About 10 30 percent of these people will go on to develop acute chest syndrome (ACS). ACS can cause further ill health. It can also cause death. Researchers want to find ways to diagnose ACS more quickly. To do this, they want to use stored blood samples and scans from a study (the DeNOVO trial) that was closed in 2015. They want to see if scans and samples taken of people with VOC who later developed ACS could help diagnose ACS faster. The data of people in the DeNOVO study who did not develop ACS will serve as controls.

Objectives:

To look at data from the DeNOVO trial to find a way to diagnose ACS more quickly.

Eligibility:

People 10 85 years old who took part in NHLBI Protocol number 05-H-0019 (the DeNOVO trial). The trial lasted from 2004 to 2008. The study was closed in November 2015.

Design:

Scans and intact, frozen samples from a study that was closed in 2015 will be studied. No new participants will be enrolled.

...

DETAILED DESCRIPTION:
Painful vasoocclusive crisis (VOC) is the most frequent acute clinical manifestation of sickle cell disease (SCD), frequently necessitating emergency department visits and/or hospitalization. Approximately 10-30% of patients admitted to the hospital with a VOC will go on to develop acute chest syndrome (ACS), a complication of SCD resulting in significant morbidity and mortality. While ACS related mortality appears to be improving in the United States, the number of hospital admissions for ACS is on the rise. Unfortunately, the diagnosis of ACS is often delayed with up to 50% of cases diagnosed two to three days after an admission for VOC. The clinical diagnosis of ACS is often delayed as it mimics other respiratory diseases. Furthermore, the lack of definitive laboratory and radiological biomarkers further confounds the ability to detect rapidly progressive ACS, a phenotype accounting for considerable ACS-related mortality. Currently, a key criterion for the diagnosis of ACS is the presence of new airspace disease on a chest radiograph in a sickle cell patient with respiratory symptoms. However, the appearance of abnormalities on chest radiography (CXR) often lags behind clinical signs and diagnostic techniques such as computed tomography (CT) which tends to reveal radiologic changes much earlier than CXR. Early diagnosis and treatment of ACS improves outcomes, hence the scientific rationale to perform such studies and develop diagnostic algorithms to facilitate early detection of ACS.

In the current study proposal, we will utilize stored blood samples and review CT scans and CXRs from 65 participants of the DeNOVO trial (NHLBI protocol # 05-H-0019). This multicenter trial conducted between 2004-08 at 11 centers including the NIH, showed that among patients with SCD hospitalized with VOC, the use of inhaled nitric oxide compared with placebo did not improve time to crisis resolution. In this study, patients enrolled at the NIH study site had baseline admission research blood drawn and thoracic CT scans performed. A repeat CT scan and repeat blood work was subsequently obtained during the development of ACS. The archived data from this subset of the study cohort therefore provides an opportunity to rigorously test the hypothesis that CT scans performed early in the setting of VOC in patients going on to develop ACS would have utility in the rapid diagnosis of this condition. Furthermore, the availability of stored plasma samples from this cohort permits the study of both imaging and plasma biomarkers in a prospectively defined sample of SCD patients. Specifically, we will identify patients admitted with VOC that went on to develop ACS and study their CT scans and plasma to determine whether these biomarkers will rapidly diagnose ACS. The patients in the same study who did not develop ACS will serve as controls.

ELIGIBILITY:
* Patients (aged 10 years and older) presenting with vaso-occlusive crisis requiring admission that were enrolled in the DeNOVO study specifically at the NIH clinical center (n=65).We will use stored blood

samples and review radiological images from these patients.

Ages: 10 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 65 participants of the DeNOVO study enrolled at the NIH
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Radiological, clinical diagnosis of Acute Chest Syndrome | 15 days from admission
  CT scans can help in the early diagnosis of acute chest syndrome.

SECONDARY OUTCOMES:
Hematological clinical diagnosis of acute chest syndrome | 15 days from admission
  sPLA2 biomarker can predict acute chest syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Arun S Shet, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States